CLINICAL TRIAL: NCT04615494
Title: Change of Internal Carotid Artery Blood Flow During Pneumoperitoneum With Steep Trendelenburg Position in Robot-Assisted Laparoscopic Prostatectomy
Brief Title: Internal Carotid Artery Blood Flow in Robot-Assisted Laparoscopic Prostatectomy
Status: Completed | Type: Observational
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Young-Kug Kim, MD, Professor, Asan Medical Center
Other Study IDs: 2020-1638
Record Dates: First submitted 2020-11-03; First posted 2020-11-04 (Actual); Last update posted 2021-01-26 (Actual); Status verified 2021-01

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Patient Positioning

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Position — Pneumoperitoneum with Steep Trendelenburg position

SUMMARY:
The purpose of this study is to evaluate the change of the internal carotid artery blood flow according to the steep trendelenburg position and pneumoperitoneum in patients undergoing robot-assisted laparoscopic prostatectomy.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have undergone robot-assisted laparoscopic prostatectomy with prostate cancer and who are 20 years or older and under 80 years
* Patients who agree to voluntarily participate in this study
* Patients with ASA class 1-2

Exclusion Criteria:

* History of diagnosis of cerebrovascular disease
* Patients who refused to participate in clinical studies

Ages: 20 Years to 79 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have undergone robot-assisted laparoscopic prostatectomy with prostate cancer
Sampling Method: Non-Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2020-11-17 (Actual); Primary Completion 2021-01-21 (Actual); Study Completion 2021-01-22 (Actual)

PRIMARY OUTCOMES:
Difference in internal carotid artery blood flow | At 10 minutes after pneumoperitoneum with steep Trendelenburg position
  Difference between the internal carotid artery blood flow measured at 10 minutes after anesthetic induction during supine position and the internal carotid artery blood flow measured at 10 minutes after pneumoperitoneum with steep Trendelenburg position

SECONDARY OUTCOMES:
Internal carotid artery blood flow | Baseline (Before anesthetic induction)
  Internal carotid artery blood flow before anesthetic induction
Internal carotid artery blood flow | At 10 minutes after anesthetic induction
  Internal carotid artery blood flow at 10 minutes after anesthetic induction
Internal carotid artery blood flow | At 10 minutes after pneumoperitoneum and Trendelenburg position
  Internal carotid artery blood flow at 10 minutes after pneumoperitoneum and Trendelenburg position
Internal carotid artery blood flow | At 30 minutes after pneumoperitoneum and Trendelenburg position
  Internal carotid artery blood flow at 30 minutes after pneumoperitoneum and Trendelenburg position
Internal carotid artery blood flow | Procedure (At skin closure)
  Internal carotid artery blood flow during supine position at skin closure

CONTACTS AND LOCATIONS:
Overall Officials: Young-Kug Kim, Professor, Study Chair — Asan Medical Center
Locations (1):
- Asan medical Center, Seoul, South Korea